CLINICAL TRIAL: NCT06188650
Title: The Efficacy and Safety of Drug Loaded Microsphere Bronchial Artery Chemoembolization (DEB-BACE) Combined With Anlotinib and Adebelimumab in the Third Line Treatment of Advanced NSCLC: a Prospective, Single Arm, Single Center, Exploratory Clinical Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ningbo Medical Center Lihuili Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2023PJ261
Record Dates: First submitted 2023-12-18; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- experimental group (Experimental)
  Interventions: Drug: Anlotinib

INTERVENTIONS:
Drug: Anlotinib — After receiving DEB-BACE treatment, the enrolled patients will rest for one week and then undergo one cycle of treatment with the combination of Anlotinib and Adebelimumab. After one course of treatment, the efficacy will be re evaluated, such as CR, and the treatment with Anlotinib and Adebelimumab will continue; For PR, SD, or PD, continue to receive DEB-BACE combined with anlotinib and adebelimumab as needed, with a maximum of 4 DEB-BACE treatments, followed by continued treatment with anlotinib and adebelimumab
  Other Names: Adebrelimab; Drug-eluting Beads Bronchial Arterial Chemoembolization，DEB-BACE

SUMMARY:
The goal of this clinical trial is to learn about Drug loaded microspheres for bronchial artery chemoembolization (DEB-BACE) combined with anlotinib and adebelimumab in patients with advanced NSCLC after second-line treatment.

The main question it aims to answer is:

The efficacy and safety of Drug Loading Beads Bronchial Arterial Chemoembolization (DEB-BACE) combined with Anlotinib and Adebelimumab in the third line treatment of advanced NSCLC.

Participants will receive DEB-BACE treatment, rest for 1 week and then undergo 1 cycle of treatment with combination of Anlotinib and Adebelimumab. With a maximum of 4 DEB-BACE treatments depending on the therapeutic effect, followed by continued treatment with Anlotinib and Adebelimumab.

ELIGIBILITY:
Inclusion Criteria:

1. Age>18 years old, gender unlimited;
2. According to the Diagnosis and Treatment Guidelines for Primary Lung Cancer (2018 Edition), NSCLC was diagnosed by pathological histology;
3. TNM staging is III - IV;
4. Failure of second-line treatment according to the CSCO guidelines;
5. ECOG PS score ≤ 2 points;
6. Estimated survival time>3 months;
7. Sign informed consent form

Exclusion Criteria:

1. Individuals who have previously received interventional therapy (iodine particle implantation, ablation, BACE treatment), or have received PD-L1 inhibitor immunotherapy during the first or second line standard treatment period of the patient;
2. Patients with other malignant tumors that have not been cured;
3. White blood cells<3 × 109/L, absolute value of neutrophils<1.5 × 109/L, neutrophil/lymphocyte ratio ≥ 3, platelet count<50 × 109/L, hemoglobin concentration<90 g/L;
4. Liver and kidney dysfunction (creatinine>176.8) μ Mol/L; Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT)>twice the normal upper limit;
5. Central squamous cell carcinoma with cavity features;
6. Incorrectable coagulation dysfunction or concomitant active massive hemoptysis;
7. Patients with concurrent active infections who require antibiotic treatment;
8. Uncontrollable hypertension, diabetes, and cardiovascular diseases with obvious symptoms;
9. Contrast agent allergy;
10. Women with concurrent pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-12-09 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
ORR | 1 year
  objective response rate

SECONDARY OUTCOMES:
PFS | 2 years
  Progression Free Survival
OS | 3 years
  Overall Survival
DCR | 3 years
  Disease Control Rate
DoR | 3 years
  Duration of Overall Response
AE | 3 years
  adverse event

CONTACTS AND LOCATIONS:
Locations (1):
- Kaitai Liu, Ningbo, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No